CLINICAL TRIAL: NCT06740292
Title: InterFlex Plate Versus Conventional Miniplates in the Management of Anterior Mandibular Fractures. a Randomized Controlled Clinical Trial
Brief Title: InterFlex Plate Versus Conventional Miniplates in the Management of Anterior Mandibular Fractures.
Acronym: InterFlex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0117-12/24
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Anterior Mandibular Fracture
Keywords: anterior mandibular fracture; symphyseal fracture; para-symphyseal fracture; InterFlex plate; functionally stabilized fixation; miniplate

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Patients were allocated in a 1:1 ratio using an on-site computer software system with concealed allocation through sequentially numbered, opaque, sealed envelopes (SNOSE). Group A was treated with InterFlex plates, and Group B with conventional miniplates
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with anterior mandibular fracture managed with conventional miniplates (Active Comparator): Patients with anterior mandibular fracture managed with conventional miniplates
  Interventions: Device: conventional miniplates
- Patients with anterior mandibular fracture managed with InterFlex plates (Experimental): Patients with anterior mandibular fracture managed with InterFlex plates
  Interventions: Device: InterFlex plates

INTERVENTIONS:
Device: conventional miniplates — conventional miniplates in double configuration
  Arms: Patients with anterior mandibular fracture managed with conventional miniplates
Device: InterFlex plates — InterFlex plates in configuration
  Arms: Patients with anterior mandibular fracture managed with InterFlex plates

SUMMARY:
the study aims to compare InterFlex plate with conventional miniplates in management of symphyseal mandibular fracture clinically regarding pain, wound healing and postoperative occlusion, and radiographically regrading bone density.

DETAILED DESCRIPTION:
A total of 18 patients with recent symphyseal mandibular fractures were allocated into two groups. Group A, comprising 9 patients, underwent treatment with the InterFlex plate, while Group B, also consisting of 9 patients, was treated with conventional two miniplates. Clinical evaluations were carried at multiple intervals up to 12 weeks postoperatively, with radiographic assessments performed immediately after surgery and at 12 weeks to measure mean bone density at the fracture line.

ELIGIBILITY:
Inclusion Criteria:

* patients with recent anterior mandibular fracture located between the mental foramina.
* adults without gender predilection who agreed to follow-up,
* fractures requiring open reduction and internal fixation, and
* those medically fit for general anesthesia were included

Exclusion Criteria:

* medically compromised patients,
* fractures with infection,
* pathological or old fractures,
* completely edentulous patients,
* comminuted fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-01-25 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Radiographic evaluation for the assessment of mean bone density at the fracture line | 3 months
  Mean bone density at the fracture line was assessed using Cone-Beam Computed Tomography (CBCT) scan in Hounsfield Units (HU)

SECONDARY OUTCOMES:
Clinical evaluation for pain | six weeks
  Pain was assessed using Visual Analogue Scale (VAS)

OTHER OUTCOMES:
Clinical evaluation for Intra-fragmentary mobility | six weeks
  Intra-fragmentary mobility was evaluated by bimanual palpation at the fracture site

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all data will be de-identified to protect the participant data. patients signed an informed consent for the use of their medical records and data for study
Supporting Information: SAP
Access Criteria: to any one who required them after deidentification